CLINICAL TRIAL: NCT06724328
Title: Maternal Heartbeat Sounds and Therapeutic Touch
Brief Title: Maternal Heartbeat Sounds and Therapeutic Touch on Heart Rate,Comfort and Behavior in Newborns
Acronym: heartbeatt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Proffesor, Pediatric Nursing Department, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DEUttouch
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Comfort; Behavior; Heart Rate
Keywords: Newborn, therapeutic touch, maternal heart, behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): In this group, preterm infants will be recorded with a camera for 20 minutes between 13:00-13:20, 19:00-19:20, and 01:00-01:20, after their routine care and feeding have been completed, with no interventions applied to the baby.
- Maternal Heartbeat (Experimental): Researchers will schedule a time with the mother within 48 hours after the baby's birth to record the heartbeat. The recording of the mother's heartbeat will be done when the mother's mood is stable and the environment is quiet. A Doppler fetal heart monitor will be used to detect the mother's heartbeat. After ensuring a regular and stable heart rate, the mother's heartbeat will be recorded for 15 minutes using a recording device.
  Interventions: Behavioral: Maternal Heartbeat
- Gentle Human Touch (Experimental): GHT will be applied to the babies at the designated times.
  Interventions: Behavioral: Gentle Human Touch
- Maternal Heartbeat and Gentle Human Touch (Experimental): For this group, maternal heartbeat will be played and GHT steps will be applied simultaneously at the designated times. Camera recording will start 2 minutes before the intervention and continue for an additional 2 minutes after the intervention.
  Interventions: Behavioral: Maternal Heartbeat and Gentle Human Touch

INTERVENTIONS:
Behavioral: Gentle Human Touch — the trained NICU nurse will place one hand's fingertips on the baby's forehead along the brow line, while the other hand will be placed around the baby's lower abdomen
  Arms: Gentle Human Touch
Behavioral: Maternal Heartbeat and Gentle Human Touch — maternal heartbeat will be played and GHT steps will be applied simultaneously at the designated times
  Arms: Maternal Heartbeat and Gentle Human Touch
Behavioral: Maternal Heartbeat — The recording of the mother's heartbeat will be done when the mother's mood is stable and the environment is quiet. A Doppler fetal heart monitor will be used to detect the mother's heartbeat. After ensuring a regular and stable heart rate, the mother's heartbeat will be recorded for 15 minutes using a recording device
  Arms: Maternal Heartbeat

SUMMARY:
This randomized controlled study aims to evaluate the effects of maternal heartbeat sounds and gentle human touch (GHT), a form of therapeutic touch, on heart rate, comfort, and behavioral scores in neonates born between 32 and 40 weeks and admitted to the neonatal intensive care unit (NICU).

DETAILED DESCRIPTION:
This parallel, randomized controlled trial will be conducted in the Neonatal Intensive Care Unit of a regional hospital. The sample will consist of 120 neonates with gestational ages of 32 to ≤40 weeks and randomly assigned to four groups (maternal heart sound, therapeutic touch, maternal heart sound + therapeutic touch, and control group). The data of the study are the Newborn Information Form, the Anderson Behavioral Status Scoring System, and Newborn Comfort Behavior Scale. Demographic data will be compared between groups (maternal heartbeat sound group (Group 1), light human touch group (Group 2), combined maternal heartbeat sound and light human touch group (Group 3), and control group (Group 4)). Video recordings will be used to compare heart rate, behavioral status, and comfort scale scores obtained before, during, and after the interventions. The time it takes to fall asleep will also be evaluated. A t-test will be applied to evaluate the score differences between groups.

ELIGIBILITY:
Inclusion Criteria:

* • Newborns between >32 and ≤40 weeks gestational age.

  * Admission to neonatal intensive care unit (NICU) after birth.
  * Parental consent form obtained.

Exclusion Criteria:

* • Absence of neurological and cardiac problems.

  * No use of corticosteroids.
  * No use of muscle relaxants.
  * Not past the postnatal 10th day.
  * Not receiving non-invasive or invasive respiratory support.

Ages: 32 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-09-03 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
comfort | 0 minutes (pre-intervention), 5 minutes, 15 minutes, and 20 minutes (post-intervention)
  It is a Likert-type scale consisting of seven parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tonus. As well as determining comfort, the COMFORTneo scale is a tool that includes numeric rating scales, which allow nurses to assess the pain and distress of the infant. The lowest score on the scale is 6, and the highest is 30. If the total score on the scale is between 14 and 30, the infant has pain or distress, is uncomfortable, and needs intervention to provide comfort. In addition, 4-6 points indicate moderate pain and distress, and 7-10 points indicate severe pain and distress

SECONDARY OUTCOMES:
behavior | 0 minutes (pre-intervention), 5 minutes, 15 minutes, and 20 minutes (post-intervention)
  It developed by Anderson et al. in 1990, evaluates the baby's sleep-wake states through 12 categories of behavioral states. ABSS involves 12 categories, including measuring the extent of eye openness, patterns of respiration, body movement, muscle tension, and crying with or without sound, to assess the behavioral state of term infants as well as premature infants.
  Categories 1-5 pertain to sleep states, 6-8 pertain to wakefulness and calmness, and 9-12 pertain to discomfort and distress. High scores indicate negative behaviors, while low scores indicate positive behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided